CLINICAL TRIAL: NCT05984953
Title: Effect of Statins and Evolocumab on Peripheral Blood Mononuclear Cell Gene Expression in Patients With Coronary Artery Disease: Yellow V
Brief Title: Rosuvastatin and Evolocumab for Coronary Artery Disease
Acronym: Yellow V
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annapoorna Kini, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-22-01743
Record Dates: First submitted 2023-04-05; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Statin: 85 patients treated with statin
  Interventions: Drug: statin
- Evolocumab: 110 patients treated with evolocumab in addition to statin or evolocumab alone
  Interventions: Drug: statin; Drug: evolocumab

INTERVENTIONS:
Drug: statin — 40 mg of rosuvastatin daily for 8-12 weeks
Drug: evolocumab — 140 mg evolocumab every 2 weeks (26 weeks)
  Groups: Evolocumab

SUMMARY:
The aim of the retrospective study is to characterize the molecular mechanisms responsible for the effect of statins and evolocumab in patients with stable coronary artery disease. The research team will retrieve and review intravascular imaging and gene expression data previously collected in the catheterization laboratory during the following time-period: 8/1/2013-4/14/2015 and 5/4/2021 - 10/28/2022.

DETAILED DESCRIPTION:
The researchers will use the previously collected transcriptomic and intravascular imaging data collected from subjects between 8/1/2013-4/14/2015 (statin group) and subjects who participated in YELLOW III study (evolocumab group). The analyses will allow us detect common and unique pathways for each drug. The researchers will use intravascular imaging findings (optical coherence tomography, OCT) to characterize patient's individual response to treatment as beneficial, if OCT fibrous cap thickness (FCT) increased at follow-up and develop machine-learning models to predict the individual response using baseline gene expression.

The researchers hypothesize that the analyses will uncover unique gene panels predicting beneficial response to statin and evolocumab allowing to select the best treatment approach for an individual patient. The total number of subjects will be 195. Transcriptomic profile of PBMC at baseline and follow-up will be compared between the groups to establish the common and distinctive molecular mechanisms of the effect of statins and evolocumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with coronary artery disease who underwent cardiac catheterization with or without PCI
* Patients from 8/1/2013-4/14/2015 and YELLOW III with both visits available, baseline and follow-up

Exclusion Criteria:

* patients from 8/1/2013-4/14/2015 and YELLOW III lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease who underwent cardiac catheterization with or without PCI
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Expression levels of mRNA in blood cells | 18 month
  Expression levels of mRNA in blood cells of the patients to be measured to identify the genes which are associated with a beneficial response to treatment using transcriptomic analysis of PBMC to find the key genes (biomarkers) responsible for effective therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  To achieve aims in the approved proposal. Proposals should be directed to annapoorna.kini@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).